CLINICAL TRIAL: NCT06903390
Title: Investigation of the Effect of Information on the Empowerment of Cancer Patients Using Question Prompt List: A Mixed Method Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Asuman Kuscu, PhD Student, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09.2022.953
Record Dates: First submitted 2025-03-19; First posted 2025-03-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms (Cancer / Tumors); Patient Participation; Patient-Centered Care; Health Communication; Patient Empowerment; Anxiety
MeSH Terms: conditions — Neoplasms; Patient Participation; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group randomized controlled trial designed to assess the impact of QPL-based communication intervention on patient empowerment and anxiety levels in cancer patients. Participants are assigned to either the intervention group (QPL-based communication) or the control group (standard physician-patient communication).
Masking Description: This study follows an open-label design, meaning that participants, care providers, and investigators are aware of the assigned intervention.
  Masking Description:
  Since this study involves a communication-based intervention, blinding is not feasible, as both participants and care providers are directly involved in delivering and receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "QPL vs. standard care to assess impact on patient empowerment & anxiety in cancer patients. (Experimental): Experimental Group 1 (QPL Communication Intervention Group) Participants in this group will receive a structured communication intervention using the Quick Question List (QPL) during their oncology examinations. The QPL aims to enhance patient empowerment, encourage active participation, and improve communication between patients and healthcare providers. It is designed to help patients express their concerns effectively and engage more actively in their care process.
  Intervention:
  Implementation of a QPL-based communication strategy in addition to standard oncology care.
  Interventions: Behavioral: QPL-based Communication Intervention
- Standard Care Group (No Intervention): Participants in this group will receive standard physician-patient communication without any additional intervention. This group serves as a control group to evaluate the effectiveness of the QPL-based communication intervention.
  Intervention:
  No additional communication tools or interventions will be applied. Patients will receive routine oncology consultations with standard physician-patient interactions.

INTERVENTIONS:
Behavioral: QPL-based Communication Intervention — This QPL-based communication intervention stands out with the following key features:
  Patient-Centered & Cancer-Specific QPL: The intervention uses a QPL tailored for cancer patients, culturally adapted to enhance empowerment and manage anxiety.
  Structured Training & Support: Patients receive training before consultations, with additional guidance for effective QPL use at subsequent visits.
  Multiple Assessment Points: The QPL's impact is measured after the first, second, and third consultations, allowing for longitudinal evaluation.
  RCT Design: This study is a randomized controlled trial (RCT), comparing the intervention group (QPL) to a control group receiving standard care.
  Focus on Empowerment & Anxiety: Unlike prior studies, this intervention focuses on empowering patients and reducing anxiety, with outcomes measured through validated scales (Patient Empowerment Scale and HADS).
  These features differentiate this intervention by offering a structured, culturally relevant approach.
  Arms: "QPL vs. standard care to assess impact on patient empowerment & anxiety in cancer patients.

SUMMARY:
Brief Summary The goal of this study is to understand how patient empowerment and a Question Prompt List (QPL) can help cancer patients.

The main questions this study aims to answer are:

What are the views of nurses, physicians, and cancer patients on patient empowerment? Does using a Question Prompt List (QPL) improve patient empowerment and reduce anxiety? Researchers will collect qualitative and quantitative data by measuring patient empowerment and anxiety levels.

Who can participate? Cancer patients receiving treatment at Private Anadolu Medical Center Hospital Nurses and physicians working with cancer patients What will participants do? Answer survey questions about their experiences with empowerment, anxiety, and communication Participate in interviews to share their thoughts on patient empowerment Use a Question Prompt List (QPL) during medical consultations Why is this study important? Many cancer patients struggle with anxiety and lack of information about their care.

A Question Prompt List (QPL) may help patients ask better questions, feel more in control of their treatment, and reduce anxiety.

This study will contribute to oncology research and help develop a culture-specific QPL for use in cancer care.

This study will take place at Private Anadolu Medical Center Hospital from January 2023 to November 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over 18 years old.
* Must understand and speak Turkish.
* Must not have any condition preventing participation (e.g., advanced dementia, cognitive impairment, speech or hearing disorders).
* For healthcare professionals in the qualitative phase: Must have at least one year of experience in oncology.

Exclusion Criteria:

* Patients without regular outpatient follow-up visits.
* Patients with severe cognitive or physiological deterioration affecting participation.
* Patients who do not comply with the study process and requirements.
* Patients who voluntarily request to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Empowerment Score | Immediately before the first consultation and within 1 day after the second and third consultations
  Assessed using the Patient Empowerment Scale to evaluate the effect of QPL-based communication on patient empowerment compared to standard communication. Higher scores indicate greater empowerment.
Change in Anxiety Level (HADS) | Immediately before the first consultation and within 1 day after the second and third consultations
  Measured using the Hospital Anxiety and Depression Scale (HADS) to assess changes in anxiety levels resulting from QPL-based communication versus standard communication. Lower scores indicate lower anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No